CLINICAL TRIAL: NCT06388941
Title: A Randomized, Controlled Study to Evaluate LNP023 (Iptacopan) in Patients With Active ANCA-associated Vasculitis
Brief Title: Iptacopan in Patients With ANCA Associated Vasculitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLNP023R12201; 2023-510525-15-00 (Other: EU CTIS)
Record Dates: First submitted 2024-04-17; First posted 2024-04-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Anti-Neutrophil Cytoplasm Antibodies (ANCA) Associated Vasculitis
Keywords: ANCA-associated vasculitis;; granulomatosis with polyangiitis (GPA);; microscopic polyangiitis (MPA);; LNP023 (iptacopan).
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis | interventions — iptacopan; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Iptacopan (Experimental): LNP023 administered orally
  Interventions: Drug: Iptacopan; Drug: Rituximab
- Control (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo; Drug: Rituximab

INTERVENTIONS:
Drug: Iptacopan — LNP023 administered orally
  Other Names: LNP023
  Arms: Iptacopan
Drug: Placebo — Matching placebo administered orally
  Arms: Control
Drug: Rituximab — Standard of care

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of iptacopan compared to standard of care (SOC) to induce and maintain remission in study participants with active granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA), when used in combination with rituximab (RTX) induction. The trial will also assess the impact of iptacopan on disease relapses, evolution of renal function and proteinuria, GC side effects, patients' immune status, and QoL.

DETAILED DESCRIPTION:
This is a randomized, controlled study to evaluate the efficacy and safety of iptacopan in combination with RTX induction therapy for the treatment of newly diagnosed or relapsed patients with active GPA or MPA.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or relapsed GPA and MPA (according to the 2022 ACR/EULAR classification criteria for GPA and MPA) requiring treatment with RTX and GC as per investigator's judgement.
* BVAS assessment with ≥1 major item, or ≥3 minor items, or ≥2 renal items at Screening.
* Positive antibody test for anti-proteinase 3 (PR3) or anti-myeloperoxidase (MPO) antibodies at Screening or with history of documented evidence of a positive antibody test.

Exclusion Criteria:

* Other systemic disease which constitutes the primary illness, including but not limited to: eosinophilic granulomatosis with polyangiitis (EGPA), moderate to severe systemic lupus erythematosus, IgA vasculitis (Purpura Schönlein-Henoch), rheumatoid vasculitis, Sjögren's syndrome, anti-glomerular basement membrane (GBM) disease, cryoglobulinemic vasculitis, autoimmune hemolytic anemia, autoimmune lymphoproliferative syndrome or mixed connective tissue disease.
* Alveolar hemorrhage requiring invasive pulmonary ventilation support at Screening.
* Severe kidney disease defined as estimated glomerular filtration rate (eGFR) <15 mL/minute/1.73m2, or kidney failure defined as receiving renal replacement therapy such as hemo(dia)filtration, hemo-/peritoneal dialysis, or having received a kidney transplant.
* Received plasma exchange/-pheresis within 12 weeks prior to Screening.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Sustained remission through Week 48 defined as complete remission at Week 24 without major relapse up to Week 48. | At Week 48
  To assess the effect of iptacopan in achieving sustained remission compared to standard of care (SOC)

SECONDARY OUTCOMES:
B cell counts | At Week 48
  To assess participant's immune status
Total IgG levels | At Week 48
  To assess participant's immune status
Complete remission at week 24 | At week 24
  Remission is defined as Birmingham Vasculitis Activity Score (BVAS) equal zero. BVAS captures various vasculitis organ manifestations as weighted score describing persistent and new symptoms with higher scores indicating more severe disease.
Time to reach BVAS=0 | At Week 24
  To assess time to remission through Week 24
Time to major relapse | At Week 48
  To assess the effect of iptacopan on disease relapse
Estimated glomerular filtration rate (eGFR) using the CKD-EPI formula, urinary protein excretion and hematuria over 48 weeks | At Week 48
  To assess the effect of iptacopan on renal function
Cumulative dose of glucocorticoid (GC) | At Week 48
  To assess the effect of iptacopan on GC sparing

CONTACTS AND LOCATIONS:
Locations (54):
- United States (4):
  - Arizona Arthritis and Rheumatology Research PLLC, Mesa, Arizona
  - UCLA Medical Center, Los Angeles, California
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Northwell Health, New York, New York
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, CABA
- Australia (4):
  - Novartis Investigative Site, Concord, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Clayton, Victoria
- Austria (3):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Leuven, Vlaams Brabant
  - Novartis Investigative Site, Roeselare, West-Vlaanderen
- Canada (4):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Fleurimont, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- China (4):
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Prague, Czechia
- Denmark (3):
  - Novartis Investigative Site, Aarhus N
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Herlev
- France (6):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (6):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Kirchheim unter Teck, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Mainz
- Hungary (3):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Novartis Investigative Site, Groningen, Netherlands
- Spain (3):
  - Novartis Investigative Site, Plasencia, Caceres
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Madrid
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Istanbul, Pendik
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
  - Novartis Investigative Site, Ankara, Yenimahalle
- United Kingdom (4):
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Brilland B, Riou J, Quemeneur T, Vandenbussche C, Merillon N, Boizard-Moracchini A, Roy M, Despre M, Piccoli GB, Djema A, Henry N, Preisser L, Blanchet O, Gnemmi V, Copin MC, Langlais D, Jeannin P, Blanco P, Delneste Y, Augusto JF; Maine-Anjou Registry Research Group. Identification of Renal Transcripts Associated with Kidney Function and Prognosis in ANCA-Associated Vasculitis. J Am Soc Nephrol. 2026 Jan 1;37(1):131-149. doi: 10.1681/ASN.0000000779. Epub 2025 Jul 9. PMID 40632630